CLINICAL TRIAL: NCT05426928
Title: Development of a Computational, Thermodynamic Model of Intraabdominal Hyperthermia in Humans Undergoing HIPEC
Brief Title: Thermodynamic Model of Hyperthermia in Humans Undergoing HIPEC
Acronym: HIPEC
Status: Recruiting | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Carlos E. Guerra, Principal Investigator, Senior Staff Anesthesiologist, Assistant Professor, Henry Ford Health System
Other Study IDs: 15538
Record Dates: First submitted 2022-06-06; First posted 2022-06-22 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: HIPEC
Keywords: Predictive model; Intraabdominal hyperthermia; Thermodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HIPEC: Adults undergoing cytoreductive surgery and who are deemed eligible for HIPEC after surgical exploration in the operating theatre.
  The patients will receive HIPEC according to routine practice, as defined by the surgical oncologist.
  Interventions: Other: Additional temperature monitoring/recording

INTERVENTIONS:
Other: Additional temperature monitoring/recording — All patients in this study will receive the same standard of care treatment for their HIPEC procedure. The only difference will be the use of additional temperature probes to collect more robust data regarding intraabdominal temperature, and the prospective collection of actual boundary conditions of the system.

SUMMARY:
Hyperthermic Intraperitoneal Chemotherapy (HIPEC) is a well-established alternative for patients with peritoneal surface malignancies. Although HIPEC has a predetermined protocol to manage body temperature, the resultant bladder and core-body temperatures are highly variable and unstable in clinical practice. Such results highlight an incomplete understanding of the thermodynamic processes during HIPEC in humans.

Previous clinical and animal investigations have studied abdominal hyperthermia, but a full human model incorporating patient variables, heat delivery, and the impact of the circulatory system and anesthesia in HIPEC has not been established.

This project seeks to develop and validate a computational thermodynamic model using prospective real-world data from humans undergoing HIPEC surgery. It is hypothesized that by incorporating patient, anesthetic, and perfusion-related variables in a thermodynamic model, the temperatures inside and outside the abdomen during HIPEC can be predicted.

DETAILED DESCRIPTION:
Peritoneal surface malignancies are a group of cancers arising from rare primary or common secondary tumors. Regardless of the etiology, the prognosis is poor and only a few therapies have shown promising results. Hyperthermic Intraperitoneal Chemotherapy (HIPEC) is a well-established alternative for patients with these malignancies. Still, as many as 46% of patients recur early after treatment.

Although HIPEC has a predetermined protocol to manage body temperature, the resultant bladder and core-body temperatures are highly variable. Age, gender, body mass index, and type and duration of chemotherapy are key factors influencing the incidence and severity of bladder hyperthermia. While clinical and animal investigations have studied abdominal hyperthermia, a full human model incorporating patient variables, heat delivery, and the impact of the circulatory system and anesthesia in HIPEC has not been established.

To bridge this gap in knowledge, this project seeks to develop and validate a computational thermodynamic model using prospective real-world data from humans undergoing HIPEC surgery. It is hypothesized that by incorporating patient, anesthetic, and perfusion-related variables in a thermodynamic model, the temperatures inside and outside the abdomen during HIPEC can be predicted. By predicting temperature changes during HIPEC, clinicians can improve the safety and efficacy of therapeutic hyperthermia.

The hypothesis will be evaluated through two specific aims:

Specific aim 1: To develop a computational, thermodynamic model of intraabdominal hyperthermia for humans undergoing HIPEC. The rationale is that existing thermodynamic models are designed for non-anesthetized or hypothermic humans, implying the need of a new model with the conditions of a HIPEC treatment.

Specific aim 2: To validate our novel computational thermodynamic model using prospective real-world data from humans undergoing HIPEC surgery. Our rationale is that by using real-world data, the initial (SA1) computational model can be optimized and ultimately used to formulate individualized hyperthermia treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adults (at least 18 years or older)
* Scheduled to undergo HIPEC surgery for abdominal cancer at HFH-Main

Exclusion Criteria:

* Pregnant females
* Minors
* Disease not amenable for treatment with HIPEC after surgical examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all patients who are scheduled to undergo hyperthermic intraperitoneal chemotherapy (HIPEC) for abdominal cancer at Henry Ford Main Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Core-body Temperature (Celsius) | Duration of HIPEC procedure (2-4 hours)
  Temperature values over time during a HIPEC treatment.
Bladder temperature (Celsius) | Duration of HIPEC procedure (2-4 hours)
  Temperature values over time during a HIPEC treatment.

SECONDARY OUTCOMES:
Mean Temperature of the Skin (C) | Duration of HIPEC procedure (2-4 hours)
  Weighed calculation of the skin temperature values over time during a HIPEC treatment.
Intrabdominal wall tissue temperature (Celsius) | Duration of HIPEC procedure (2-4 hours)
  Temperature values over time during a HIPEC treatment.
Set Temperature (Celsius) | Duration of HIPEC procedure (2-4 hours)
  Temperature values over time during a HIPEC treatment
Inflow Temperature (Celsius) | Duration of HIPEC procedure (2-4 hrs)
  Temperature values over time during a HIPEC treatment
Outflow Temperature (Celsius) | Duration of HIPEC procedure (2-4 hours)
  Temperature values over time during a HIPEC treatment
HIPEC Flow | Duration of HIPEC procedure (2-4 hours)
  Flow values (mL/min) over time during a HIPEC treatment
Operating Room Temperature (Celsius) | Duration of HIPEC procedure (2-4 hours)
  Temperature values over time during a HIPEC treatment
Underbody Blanket Temperature (Celsius) | Duration of HIPEC procedure (2-4 hours)
  Temperature values over time during a HIPEC treatment
Convection Air Blanket Temperature (Celsius) | Duration of HIPEC procedure (2-4 hours)
  Temperature values over time during a HIPEC treatment
Intrabdominal Cavity Volume (mL) | Preoperative, on average within 3 months prior to surgery.
  3D-lab post-processing of preoperative CT scans.
Peritoneal Cavity Volume (mL) | Preoperative, on average within 3 months prior to surgery.
  3D-lab post-processing of preoperative CT scans.
Abdominal Volume (mL) | Preoperative, on average within 3 months prior to surgery.
  3D-lab post-processing of preoperative CT scans.
Blood Pressure (mmHg) | Duration of HIPEC procedure (2-4 hours)
  Blood pressure values over time during a HIPEC treatment.
Heart Rate (beats/min) | Duration of HIPEC procedure (2-4 hours)
  Heart rate values over time during a HIPEC treatment.
Cardiac Output (L/min) | Duration of HIPEC procedure (2-4 hours)
  Cardiac output values over time during a HIPEC treatment.
Stroke Volume Variation (%) | Duration of HIPEC procedure (2-4 hours)
  Stroke volume variation values over time during a HIPEC treatment.
Body fat percentage (%) | Preoperative, obtained the day of surgery.
  Determined by impedancemetry
Weight (Kg) | Preoperative, obtained the day of surgery.
  Participant's weight
Height (m) | Preoperative, obtained the day of surgery.
  Participant's height

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Guerra, MD, Principal Investigator — Staff Anesthesiologist
Locations (1):
- Katherine Nowak, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Loke DR, Helderman RFCPA, Rodermond HM, Tanis PJ, Streekstra GJ, Franken NAP, Oei AL, Crezee J, Kok HP. Demonstration of treatment planning software for hyperthermic intraperitoneal chemotherapy in a rat model. Int J Hyperthermia. 2021;38(1):38-54. doi: 10.1080/02656736.2020.1852324. PMID 33487083
- [Background] Ladhari T, Szafnicki K. Modelling of some aspects of a biomedical process: application to the treatment of digestive cancer (HIPEC). 3 Biotech. 2018 Apr;8(4):190. doi: 10.1007/s13205-018-1211-5. Epub 2018 Mar 20. PMID 29564201
- [Background] Stolwijk JA, Nadel ER, Wenger CB, Roberts MF. Development and application of a mathematical model of human thermoregulation. Arch Sci Physiol (Paris). 1973;27(3):303-10. No abstract available. PMID 4807388
- [Background] Severens NM, van Marken Lichtenbelt WD, Frijns AJ, Van Steenhoven AA, de Mol BA, Sessler DI. A model to predict patient temperature during cardiac surgery. Phys Med Biol. 2007 Sep 7;52(17):5131-45. doi: 10.1088/0031-9155/52/17/002. Epub 2007 Aug 7. PMID 17762076